CLINICAL TRIAL: NCT06138197
Title: Comparative Evaluation of Three Surgical Robotic Platforms for the Laparoscopic Hysterectomy Procedure: Post Market Clinical Follow Up Study
Brief Title: Comparison of Three Robotic Platforms for Hysterectomy
Acronym: COMPAR-HYST
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Clinical Professor, Universita di Verona
Other Study IDs: COMPAR-HYST
Record Dates: First submitted 2023-04-01; First posted 2023-11-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; Gynecologic pathology; Robotic-assisted laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Robotic-assisted hysterectomy by da Vinci X surgical system, model IS4200 (INTUITIVE): Women who undergo robotic-assisted hysterectomy by da Vinci X surgical system, model IS4200 (INTUITIVE)
  Interventions: Procedure: Robotic-assisted hysterectomy
- Robotic-assisted hysterectomy by VERSIUS ® surgical system (ROBOTIC SURGICAL SYSTEM): Women who undergo robotic-assisted hysterectomy by VERSIUS ® surgical system (ROBOTIC SURGICAL SYSTEM)
  Interventions: Procedure: Robotic-assisted hysterectomy
- Robotic-assisted hysterectomy by HUGO ™ Robotic Assisted Surgery System (RAS) (MEDTRONIC): Women who undergo robotic-assisted hysterectomy by HUGO ™ Robotic Assisted Surgery System (RAS) (MEDTRONIC)
  Interventions: Procedure: Robotic-assisted hysterectomy

INTERVENTIONS:
Procedure: Robotic-assisted hysterectomy — Robotic-assisted hysterectomy following usual surgical technique

SUMMARY:
Hysterectomy is the most common procedure in gynaecology after a cesarean section. In recent years, the laparoscopic approach has become preferred given the different advantages over the traditional laparotomic approach, and both conventional laparoscopy and robotic-assisted laparoscopy have become the standard approach for hysterectomy. To date, robotic-assisted laparoscopic hysterectomy has been performed using one robotic platform and only recently, two new robotic platforms have been introduced in clinical practice. Although all three are registered for human use and available for clinical practice, there are currently not enough clinical experiences and data in the literature to evaluate the efficacy, safety and relationship between cost and efficacy of the new platforms available for the robotic-assisted laparoscopic hysterectomy. For this reason, the investigators will conduct an exploratory clinical study on a Post Market Clinical Follow up (PMCF) medical device aimed at performing a preliminary assessment of the global performance of the ITL procedure implemented using the three robotic platforms currently available.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total laparoscopic hysterectomy surgery
* Age > 18 years
* Signature of the informed consent

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients who are candidates for hysterectomy for a non-gynaecological indication
* Patients undergoing previous radiation therapy
* Patients unable to express adequate informed consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women undergoing robotic-assisted elective total laparoscopic hysterectomy
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Textbook outcome satisfaction | 90 days after surgery
  Robotic-assisted hysterectomy performed without laparotomy conversion, intraoperative complications, postoperative complications (Clavien-Dindo classification ≥2), the performance of postoperative imaging excluding transvaginal ultrasound, reoperation, length of stay after day of surgery >2 days, readmission within 90 days, mortality, surgery length greater than 120 minutes, or intraoperative blood loss greater than 100mL. The Textbook outcome will be considered fulfilled if all conditions are met.

SECONDARY OUTCOMES:
Intraoperative complications | During surgery
  Intraoperative complications graded based on the Clavien-Dindo classification
Postoperative complications | 30 and 90 days after surgery
  Postoperative complications graded based on the Clavien-Dindo classification
Operative time | During surgery
  Time between first incision and skin closure
Intraoperative blood loss | During surgery
  Total blood aspirate during the surgical procedure
Sexual function | 90 and 180 days after surgery
  The female sexual function index (FSFI) consists of 19 multiple-choice items that assess female sexual functioning based on 6 domains: desire, arousal, orgasm, pain, sexual satisfaction, and lubrication. The total score ranges from 0 to 36, with 26.55 as the cut-off suggesting the presence of sexual dysfunction. The higher the score, the better the sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Principal Investigator — Universita di Verona; Simone Garzon, MD, Principal Investigator — Universita di Verona; Pier Carlo Zorzato, MD, Principal Investigator — Universita di Verona
Locations (1):
- AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torpy JM, Lynm C, Glass RM. JAMA patient page. Hysterectomy. JAMA. 2004 Mar 24;291(12):1526. doi: 10.1001/jama.291.12.1526. No abstract available. PMID 15039420
- [Background] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Background] Lawrie TA, Liu H, Lu D, Dowswell T, Song H, Wang L, Shi G. Robot-assisted surgery in gynaecology. Cochrane Database Syst Rev. 2019 Apr 15;4(4):CD011422. doi: 10.1002/14651858.CD011422.pub2. PMID 30985921
- [Background] Nobbenhuis MAE, Gul N, Barton-Smith P, O'Sullivan O, Moss E, Ind TEJ; Royal College of Obstetricians and Gynaecologists. Robotic surgery in gynaecology: Scientific Impact Paper No. 71 (July 2022). BJOG. 2023 Jan;130(1):e1-e8. doi: 10.1111/1471-0528.17242. Epub 2022 Jul 17. PMID 35844092
- [Background] Monterossi G, Pedone Anchora L, Gueli Alletti S, Fagotti A, Fanfani F, Scambia G. The first European gynaecological procedure with the new surgical robot Hugo RAS. A total hysterectomy and salpingo-oophorectomy in a woman affected by BRCA-1 mutation. Facts Views Vis Obgyn. 2022 Mar;14(1):91-94. doi: 10.52054/FVVO.14.1.014. PMID 35373554